CLINICAL TRIAL: NCT02474940
Title: Enhancing the Benefits of Pain and Fatigue Treatment in MS
Brief Title: MS Symptom Management Study
Acronym: ENHANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Mark Jensen, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 46765-EB; RG 5232-A-4 (Other Grant/Funding Number: National Multiple Sclerosis Society)
Record Dates: First submitted 2015-05-21; First posted 2015-06-18 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Multiple Sclerosis; Chronic Pain; Fatigue
Keywords: Multiple Sclerosis; Chronic Pain; Chronic Fatigue; Autoimmune Diseases; Autoimmune Diseases of the Nervous System; Central Nervous System Diseases; Demyelinating Autoimmune Diseases, CNS; Demyelinating Diseases
MeSH Terms: conditions — Multiple Sclerosis; Chronic Pain; Fatigue; Autoimmune Diseases; Autoimmune Diseases of the Nervous System; Central Nervous System Diseases; Demyelinating Autoimmune Diseases, CNS; Demyelinating Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention #1 (Experimental): NF-HYP
  Interventions: Behavioral: Intervention #1
- Intervention #2 (Experimental): MM-HYP
  Interventions: Behavioral: Intervention #2
- Intervention #3 (Experimental): HYP-ONLY
  Interventions: Behavioral: Intervention #3

INTERVENTIONS:
Behavioral: Intervention #1 — Intervention #1 consists of 11 treatment sessions over 6-12 weeks (1-2 sessions/week on average). Sessions 1-6 will involve neurofeedback training. During neurofeedback training, sensors will be placed on a subject's head and ears, and s/he will be able to hear sounds on a computer that correspond to his/her brainwaves. The subject will learn how to change his/her brainwaves by changing the sounds heard. Session 7 will be a face-to-face self-hypnosis session. During self-hypnosis training, subjects will learn to enter a state of focused attention, and then change how he/she experiences pain and/or fatigue. In sessions 8-11, subjects will listen to an audio recording of a self-hypnosis training session. Subjects will complete one neurofeedback training session immediately before each of these four hypnosis sessions. A relaxation and hypnotic exercise will also be done during two of the 11 sessions.
  Arms: Intervention #1
Behavioral: Intervention #2 — Intervention #2 consists of 11 treatment sessions over 6-12 weeks (1-2 sessions/week on average). Sessions 1-6 will involve mindfulness meditation training. During mindfulness training, subjects will be asked to focus their attention on an object of awareness, such as their breath. Subjects will then be asked to focus on their feelings/thoughts during the training. Session 7 will be a face-to-face self-hypnosis session. During self-hypnosis training, subjects will learn to enter a state of focused attention, and then change how he/she experiences pain and/or fatigue. In sessions 8-11, subjects will listen to an audio recording of a self-hypnosis training session. Subjects will complete one mindfulness meditation training session immediately before each of these four hypnosis sessions. A relaxation and hypnotic exercise will be done during two of the 11 sessions. On three of the 11 sessions, research staff will also place sensors on a subject's head and ears to measure brainwaves.
  Arms: Intervention #2
Behavioral: Intervention #3 — Intervention #3 consists of five treatment sessions of self-hypnosis training during the treatment phase of the study (1-2 sessions/week on average). The treatment phase of the study will last about 6-12 weeks. During the first 4-5 weeks, subjects in Intervention #3 will not be asked by study researchers to do anything. At the end of this waiting period, subjects will complete a set of telephone interviews. Subjects will then attend one face-to-face self-hypnosis training session. During self-hypnosis training, subjects will learn to enter a state of focused attention, and then change how he/she experiences pain and/or fatigue. In the last four sessions, subjects will listen to an audio recording of a self-hypnosis training session. A relaxation and hypnotic exercise will also be done during two of the five sessions.
  Arms: Intervention #3

SUMMARY:
People with Multiple Sclerosis (MS) often have pain and/or fatigue. Unfortunately, available treatments provide inadequate relief for the majority of these individuals. There remains an urgent need for additional treatment options for MS-related symptoms. The purpose of this study is to see if alternative treatments that involve self-hypnosis training, neurofeedback training and/or mindfulness meditation training, or a combination of some of these treatments can help decrease pain and fatigue in people with MS. A subject must have a diagnosis of MS, have chronic pain and/or fatigue, and be at least 18 years old to participate, among other criteria.

DETAILED DESCRIPTION:
Individuals from the study's recruitment sources with an MS diagnosis will be contacted by research staff via telephone and invited to be screened for participation. In addition, individuals interested in participating may contact research staff upon learning about the study through a description listed on an approved website, flyer, or a referral. Research staff will use a recruitment script for purposes of screening subjects and explaining the study. In addition, the initial screening process will also include a 6-item cognitive screening and a psychological screening assessment done by a licensed clinician.

Research staff will verify the MS diagnosis of prospective subjects who have not been 'pre-verified' in one of three ways during the recruitment process:

1. Research staff will attempt to determine whether a subject has a University of Washington Medical Center (UWMC) or Harborview Medical Center (HMC) medical record by conducting a simple search using a secure application.

   If research staff are unable to locate a medical record for the prospective subject, or if the individual contacts research staff after seeing the study description on an approved website or flyer, then one of two options will be pursued:
2. Subjects will be asked during the initial screening process if staff may review their medical records if they have received services at the UWMC/HMC since their diagnosis;
3. Subjects will be asked during the initial screening process if staff may contact a physician of their choice to verify their diagnosis if (a) they have not received services at the UWMC/HMC since their diagnosis; (b) they refuse to give staff permission to review their UWMC/HMC medical records; or (c) staff for some reason cannot find a UWMC/HMC medical record despite the subject attesting to being a patient at one time at the UWMC/HMC and giving staff permission to review his/her records.

Only individuals whose diagnosis has been verified (either via medical record review prior to/during screening or through verification via the subject's physician depending on recruitment source) will proceed with the psychological screening assessment.

Once a prospective subject has been screened as eligible and gotten their MS diagnosis verified, research staff will arrange a time and date for the prospective subject to participate in a telephone psychological screening assessment with one of the study's licensed clinicians. The study clinician will ask potential subjects some questions to assess the presence of active suicidal ideation or paranoid thoughts using an assessment sheet. Individuals who do have these types of thoughts will not be eligible for the study. Individuals will be referred to a mental health professional if he or she needs immediate attention.

Research staff will then arrange a time with the subject to attend an in-person initial intake session. At the beginning of the initial intake session, research staff will review a consent form with the subject and answer any questions he/she may have. The subject will complete and sign the consent form if he/she would like to participate. If the subject decides to enroll in the study, he/she will then be asked to participate in a relaxation and hypnotic exercise, and provide basic demographic and contact information, as well as information about their MS diagnosis and pain and/or fatigue problem(s) he/she experiences. The initial intake session will last about 1.5 hours depending on the subject's answers.

Subjects will be randomly assigned (by chance, like flipping a coin) to one of three treatment interventions. All three treatment interventions involve learning self-hypnosis techniques. During self-hypnosis, subjects learn to enter a state of focused attention, and then change how they experience pain and/or fatigue. Two of the three treatment interventions will also include mindfulness meditation or neurofeedback training. Investigators are interested in comparing the three different approaches to treating chronic pain and/or fatigue.

A research staff member will also contact each subject four times by telephone during his/her participation in the study to complete three short interviews or assessments, 3-5 minutes long, and one longer assessment, about 30-40 minutes long, in a period of one week. These assessments will be completed one week prior to the treatment period, about halfway through the treatment period, after the completion of treatment, and 1-month after the subject completes treatment. The three shorter assessments will include questions about pain intensity. The fourth longer assessment will include questions about such things as how the subject thinks about pain and fatigue, treatments for pain and/or fatigue the subject has received, medications or drugs the subject has used, and any depressive symptoms the subject may have experienced.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of MS
* Moderate to severe chronic pain and/or fatigue
* Able to read, speak, and understand English

Exclusion Criteria:

* Severe cognitive impairment defined as two or more errors on the Six-Item Screener
* History of seizure activity
* Psychiatric condition or symptoms that would interfere with participation
* Currently receiving psychological treatment for pain and/or fatigue
* Has participated in any previous or current research study conducted by investigators in the Department of Rehabilitation Medicine that involved pain or fatigue management via psychological treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in average pain intensity pre-treatment to post-treatment | Pre-treatment (1 week before Session 1), Mid-treatment (1 week before Session 7), Post-treatment (within a week after Session 11), 1-month following end of treatment
  Average pain intensity will be assessed via telephone interviews using a 0-10 numerical rating scale (NRS) of average pain in the past 24 hours, four times within a 1-week period at each assessment point.
Change in average fatigue severity pre-treatment to post-treatment | Pre-treatment (1 week before Session 1), Mid-treatment (1 week before Session 7), Post-treatment (within a week after Session 11), 1-month following end of treatment
  Fatigue severity will be assessed with the Fatigue Severity Scale (FSS). The 9-item FSS asks respondents to rate fatigue and the extent to which it interferes with activities on 1 (Strongly disagree) to 7 (Strongly agree) scales. The FSS is assessed once at each assessment point.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jensen, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Ninth and Jefferson Building, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No